CLINICAL TRIAL: NCT04078698
Title: Documentation of the Safety and Effectiveness Profile of the IgG Immunoadsorber GLOBAFFIN® in Clinical Routine (SEPIAR)
Brief Title: Documentation of the Safety and Effectiveness Profile of the IgG Immunoadsorber GLOBAFFIN® in Clinical Routine
Acronym: SEPIAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Alcedis GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TA-IA-03-INT
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Autoimmune Diseases
Keywords: Therapeutic apheresis; Immune apheresis
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Intervention Model Description: Prospective, multi-centre, open-label, non-comparative, interventional study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with the IgG immunoadsorber GLOBAFFIN® (Experimental): Treatment with the IgG immunoadsorber GLOBAFFIN® in clinical routine according to their intended use.
  Interventions: Device: Immunoadsorber GLOBAFFIN®

INTERVENTIONS:
Device: Immunoadsorber GLOBAFFIN® — Documentation of the treatment with one of the immunoadsorber GLOBAFFIN® depending on the patient's underlying disease

SUMMARY:
Documentation of the safety and effectiveness profile of the CE-labelled immunoadsorber GLOBAFFIN® in clinical routine according to their intended use.

DETAILED DESCRIPTION:
The objective of the study is the documentation of the safety and effectiveness profile of the CE-labeled immunoadsorber GLOBAFFIN® in clinical routine according to their intended use.

The primary objective for the IgG adsorber GLOBAFFIN® is the estimation of the mean relative reduction in total IgG from pre- to post-treatment per treatment session.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years
* Informed consent signed and dated by study patient and investigator/authorised physician
* Ability to understand the nature and requirements of the study
* Treatment with one of the immunoadsorber system GLOBAFFIN® according to the intended use.

Exclusion Criteria:

General:

* Any condition which could interfere with the patient's ability to comply with the study
* In case of female patients: pregnancy or lactation period (if patient is ≥ 55 years old or have been surgically sterilized, a negative pregnancy test is not required)
* Participation in an interventional clinical study during the preceding 30 days.
* Participation in an interventional clinical study with pharmacological active substances (e.g. therapeutic antibodies) during the preceding 60 days.
* Any deviation from the intended use

Study-specific:

Any contraindication listed in the valid instruction for use:

* Hypersensitivity or allergy against any materials used in either the immunoadsorber column or the extracorporeal circuit
* Inability to withstand the stress of an extracorporeal treatment procedure due to their age, their physical developments or their clinical constitution
* Previously demonstrated hypersensitivity associated with therapeutic apheresis
* No suitable anticoagulation treatment, such as due to known hypersensitivity to heparin or ACD-A
* Haemorrhagic diathesis in which extracorporeal apheresis procedures and anticoagulation performed have a high bleeding hazard
* Severe cardiovascular disease, so that extracorporeal treatment is not possible
* Acute, systemic infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-08-15 (Actual)

PRIMARY OUTCOMES:
Relative reduction in total IgG from pre- to post-treatment for GLOBAFFIN® | 5 years

SECONDARY OUTCOMES:
Mean relative reduction in disease-specific IgG, total IgM and total IgA | 5 years
Clinical effect of the treatment measured by the physician's judgement as well as indication specific scores | 5 years

OTHER OUTCOMES:
Adverse events and serious adverse events during the treatment, reported incidents, device deficiencies and handling problems | 5 years
Reduction of laboratory safety parameters | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan T. Kielstein, Prof. Dr., Principal Investigator — Academic Teaching Hospital Braunschweig
Locations (3):
- Germany (3):
  - Städtisches Klinikum Braunschweig, Braunschweig, Lower Saxony
  - Diakonissenkrankenhaus Flensburg, Flensburg
  - University of Ulm - Department of Neurology, Ulm